CLINICAL TRIAL: NCT06964932
Title: Efficacy and Safety of Pasteurized Akkermansia Muciniphila Akk11 in Obesity/Overweight Weight Management and Energy Metabolism:a Randomized, Double-blind, Placebo-controlled Trial
Brief Title: Probiotics in Obesity Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wecare Probiotics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WK20250424
Record Dates: First submitted 2025-04-22; First posted 2025-05-11 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic group (Experimental): Pasteurized Akkermansia muciniphila Akk11 capsule, 100 billion TFU/day
  Interventions: Dietary Supplement: Probiotc
- Placebo group (Placebo Comparator): Placebo capsule, one capsule/day
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotc — The trial phase of this study lasted 12 weeks, and each patient will make 4 visits (week 0, week 4, week 8， week 12)
  Arms: Probiotic group
Dietary Supplement: Placebo — The trial phase of this study lasted 12 weeks, and each patient will make 4 visits (week 0, week 4, week 8， week 12)
  Arms: Placebo group

SUMMARY:
Evaluate the effects of pasteurized Akkermansia muciniphila Akk11 (killed bacteria) capsules compared to placebo on body composition parameters (including weight, BMI, body fat percentage, waist - hip ratio (WHR), wrist circumference, visceral fat area, and basal metabolic rate) and blood lipid levels (total cholesterol (TC), low - density lipoprotein (LDL), high - density lipoprotein (HDL), and triglycerides (TG)) in overweight or obese adults.

ELIGIBILITY:
Inclusion Criteria:

1. A body mass index (BMI) of 24 kg/m² or above;
2. Voluntarily signing an informed consent form to take part in the study;
3. Willingness to undertake the study protocol and associated restrictions, such as adhering to a calorie - restricted - low carbohydrate diet;
4. No intention to become pregnant from 14 days before screening, and commitment to using effective contraception until six months after the trial concludes.

Exclusion Criteria:

1. Intake of products akin to the test product in the recent period that might sway the outcomes;
2. Presence of mental or neurological disorders, celiac disease, lactose intolerance, or allergic conditions;
3. Being pregnant, breastfeeding, or planning to conceive;
4. Past diagnosis of Irritable Bowel Syndrome, Ulcerative Colitis, Hepatic Cirrhosis, or Diabetes Mellitus;
5. Use of antibiotics in the preceding three months;
6. Inability to comply with the test product regimen or attend follow-up visits regularly, making efficacy assessment unfeasible;
7. Smoking in excess of 10 cigarettes daily;
8. Hypersensitivity to probiotic products;
9. Any other participants deemed unsuitable for the research by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2025-03-15 (Actual); Primary Completion 2025-12-03 (Actual); Study Completion 2026-01-28 (Actual)

PRIMARY OUTCOMES:
Change in body weight before and after intervention | Week 0 , Week 4, Week 8, Week 12
  Measured using a calibrated scale

CONTACTS AND LOCATIONS:
Locations (1):
- The School of Food and Bioengineering, Henan University of Science and Technolog, Luoyang, Henan, China